CLINICAL TRIAL: NCT04643587
Title: A Phase 1, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Exploratory Efficacy of Nebulized CSL787 in Healthy Subjects and Subjects With Non-Cystic Fibrosis Bronchiectasis (NCFB)
Brief Title: Study to Assess CSL787 in Non-cystic Fibrosis Bronchiectasis (NCFB)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSL787_1001; 2020-002684-66 (EudraCT Number)
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Noncystic Fibrosis Bronchiectasis (NCFB)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- CSL787 (SAD dose 1) (Experimental): Inhalation by mouth of a nebulized aerosol in healthy subjects
  Interventions: Biological: CSL787
- CSL787 (SAD dose 2) (Experimental): Inhalation by mouth of a nebulized aerosol in healthy subjects
  Interventions: Biological: CSL787
- CSL787 (SAD dose 3) (Experimental): Inhalation by mouth of a nebulized aerosol in healthy subjects
  Interventions: Biological: CSL787
- CSL787 (SAD dose 4) (Experimental): Inhalation by mouth of a nebulized aerosol in healthy subjects
  Interventions: Biological: CSL787
- CSL787 (MAD dose 1) (Experimental): Inhalation by mouth of a nebulized aerosol in NCFB subjects
  Interventions: Biological: CSL787
- CSL787 (MAD dose 2) (Experimental): Inhalation by mouth of a nebulized aerosol in NCFB subjects
  Interventions: Biological: CSL787
- CSL787 (MAD dose 3) (Experimental): Inhalation by mouth of a nebulized aerosol in NCFB subjects
  Interventions: Biological: CSL787
- Placebo (Placebo Comparator): Inhalation by mouth of a nebulized aerosol
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSL787 — Human plasma-derived polyvalent immunoglobulin G (IgG) administered via inhalation of an aerosol produced using a nebulizer
  Arms: CSL787 (MAD dose 1); CSL787 (MAD dose 2); CSL787 (MAD dose 3); CSL787 (SAD dose 1); CSL787 (SAD dose 2); CSL787 (SAD dose 3); CSL787 (SAD dose 4)
Drug: Placebo — Normal saline (0.9% NaCl)
  Arms: Placebo

SUMMARY:
This study is a prospective, multicenter, randomized, double-blind, placebo-controlled study to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and exploratory efficacy of nebulized CSL787 after administrations of single (SAD) ascending doses in healthy subjects and multiple (MAD) ascending doses in subjects with NCFB.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years at the time of providing written informed consent

For Part A (SAD) Only:

* Healthy and free of medical conditions that could in the opinion of the investigator affect's the subject's participation in the study or the interpretation of results.

For Part B (MAD) Only:

* Diagnosis of NCFB made by a respiratory physician, confirmed per CT showing bronchial wall dilatation with or without bronchial wall thickening, with a FEV1 ≥ 40% of the predicted value regarding age, height, gender, ethnicity, and FEV1 ≥ 1 L (pre-bronchodilator values) at the Screening Visit.
* No antibiotic use within 1 month before the Screening Visit.
* Presence of one or more of the following bacteria (H. influenzae, P. aeruginosa, M. catarrhalis, S. pneumoniae, members of Enterobacterales family or S. aureus) in the sputum culture at the Screening Visit.
* Has been fully vaccinated against COVID-19 (as per country recommendations) at least 7 days prior to Day 1

Exclusion Criteria:

* Evidence of a clinically significant medical condition, disorder, or disease, including but not limited to any of the following: hepatic (hepatitis, cirrhosis); biliary; renal; cardiac; bronchopulmonary; vascular; hematologic; gastrointestinal; allergy; endocrine / metabolic (diabetes, thyroid disorders, adrenal disease); neurologic; psychiatric; immunodeficiency; cancer.
* History of chronic respiratory disease (eg, COPD or bronchiectasis) or current asthma with regular treatment including occasional use of an inhaler for exercise induced asthma.
* Current moderate-severe allergic disease (eg, allergic rhinitis) with regular treatment.
* Diagnosis of cystic fibrosis, mycobacterial disease, connective tissue disease, or alpha-1 antitrypsin deficiency as underlying disease for bronchiectasis.
* Oral/parenteral corticosteroid 28 days before the Screening Visit until EOS Visit. Use of long acting bronchodilators (long acting muscarinic antagonists (LAMA) and / or long acting beta2 agonists (LABA) and/or inhaled corticosteroids that have been at a stable dose for at least 3 months before the Screening Visit is permitted; inhalation with hypertonic saline solution is permitted up to and including Day -1.
* Any systemic or inhaled antibiotic for acute pulmonary exacerbation within 1 month before the Screening Visit until EOS Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment emergent adverse events (TEAEs) - overall, severity and causality | Up to 8 days (healthy volunteers); Up to 21 days (NCFB patients)
Percent of subjects with TEAEs - overall, severity and causality | Up to 8 days (healthy volunteers); Up to 21 days (NCFB patients)

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of CSL787 in sputum and serum in healthy subjects | Up to 8 days from inhalation
Time of maximum concentration (Tmax) of CSL787 in sputum and serum in healthy subjects | Up to 8 days from inhalation
Area under the concentration-time curve from time 0 to 24 hours (AUC0-24h) of CSL787 in sputum and serum in healthy subjects | Up to 8 days from inhalation
Area under the concentration-time curve from time 0 to last quantifiable time point (AUC0-last) of CSL787 in sputum and serum in healthy subjects | Up to 8 days from inhalation
Area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) of CSL787 in sputum and serum in healthy subjects | Up to 8 days from inhalation
Apparent total clearance of the drug (CL/F) of CSL787 in sputum and serum in healthy subjects | Up to 8 days from inhalation
Apparent volume of distribution during the elimination phase (V/F) of CSL787 in sputum and serum in healthy subjects | Up to 8 days from inhalation
Terminal elimination half-life (T1/2) of CSL787 in sputum and serum in healthy subjects | Up to 8 days from inhalation
Cmax of CSL787 in sputum and serum of NCFB subjects | On Day 1, after dosing
Tmax of CSL787 in sputum and serum of NCFB subjects | On Day 1, after dosing
Ctrough of CSL787 in sputum and serum of NCFB subjects | On Day 1, after dosing
AUCtau of CSL787 in sputum and serum of NCFB subjects | On Day 1, after dosing
Cmax of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
Tmax of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
Ctrough of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
AUCtau of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
T1/2 of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
CL/F of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
V/F of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
Accumulation Ratio (AR) for Cmax of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
AR for Ctrough of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose
AR for AUCtau of CSL787 in sputum and serum of NCFB subjects | On Day 14, after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (3):
- IKF Pneumologie Institute, Frankfurt, Germany
- United Kingdom (2):
  - Medicines Evaluation Unit (MEU), Manchester, England
  - Celerion, Belfast, Northern Ireland

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.